CLINICAL TRIAL: NCT07255664
Title: A FIH, Phase I/IIa, Open-label Trial Assessing Safety, Tolerability, and Feasibility of Repeated Administrations of a Novel Autologous TIL-based Immunotherapy in Patients With Metastatic Colorectal or Prostate Cancer
Brief Title: A FIH, Phase I/IIa, Trial Assessing Feasibility of Administrations of TIL-based Immunotherapy in Patients With Metastatic CRC and PC
Acronym: ProbeTILity
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Curacell Holding AB (Industry)
Collaborators: Zellwerk GmbH (Unknown); Frankfurter Institut für Klinische Krebsforschung IKF GmbH (Unknown); Krebsforschung Rhein-Main e.V. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CuraCell-Ger-01; 2025-521227-70-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Cancer; Prostate Cancer Metastatic; Prostate Cancer Locally Advanced
Keywords: mCRC; aPC; TIL; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab; Cyclophosphamide; Interleukin-2; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CC-38 Drug Product (Experimental): The advanced therapy investigational medicinal product (ATIMP) of this trial is an autologous tumor infiltrating lymphocytes (TIL)/ personalized TIL administration (product name CC-38).
  Interventions: Drug: CC-38; Drug: Pembrolizumab; Drug: Cyclophosphamid; Drug: Interleukin-2; Drug: Uromitexan

INTERVENTIONS:
Drug: CC-38 — CC-38 drug product is an autologous ATIMP composed of in vitro expanded tumor-infiltrating T-lymphocytes.
Drug: Pembrolizumab — A concomitant IMP is pembrolizumab
  Other Names: Keytruda
Drug: Cyclophosphamid — Cyclophosphamid is used as a AxMP
Drug: Interleukin-2 — Interleukin-2 is used as a AxMP.
  Other Names: Proleukin S
Drug: Uromitexan — Uromitexan is used as a AxMP.

SUMMARY:
This is a First-In-Human trial investigating a novel expansion protocol of an ATIMP (CC-38), composed of autologous TIL.

DETAILED DESCRIPTION:
T-cell therapies have demonstrated successful responses in solid tumors, most frequently studied in malignant melanomas. In the present trial, we include patients with metastatic colorectal cancer and metastatic prostate cancer, two cancer forms that have not been well studied in T-cell therapy studies, yet.

In the ProbeTILity trial we hypothesize that in patients with metastatic CRC or metastatic prostate cancer ex vivo expansion of repeated re-administration of TIL establishes a more long-term persistence of TILS in the patient´s blood stream, that could increase the likelihood of tumor infiltration by TILs.

ELIGIBILITY:
Inclusion Criteria:

* Patient (female or male) has signed informed consent according to ICH/GCP and national/local regulations prior to any trial-specific procedure.
* Patient is 18 years or older at the time of signing the informed consent form.
* Patient must live in an area where a hospital for care can be reached within a maximum of 50 km.
* Patient has histological or cytological confirmation of:

  * colorectal cancer, which is stage IV (any T / any N / M1), not amenable to curative surgery, OR
  * prostate cancer, which is stage III locally advanced, not amenable to curative surgery (T3-4 / N0 / M0 or any T / N1 / M0), or stage IV metastatic (any T / any N / M1)
* Patient has received all lines of therapy that

  * are considered SOC for the patient's indication according to applicable European/national professional society medical guidelines and local medical practice at time of enrollment
  * are available via the national health insurance system and the patient is considered eligible for but led to insufficient response or were medically not justified or refused by the patient.
* Patient has confirmed disease progression by radiologic imaging from the previous line of therapy.
* Patient has sufficient amount of previously not irradiated tumor tissue in adequate quality for TIL harvest and expansion, i.e., either:

  * Primary or metastatic lesion has been selected for surgery (e.g., to reduce tumor burden, pain relief), Or
  * Patient has consented to surgery for the purpose of tissue harvesting for TIL expansion and is considered suitable to undergo surgery for this purpose. Note: Patients with a non-justifiable anesthesiologic and/or surgical risk, as determined by the investigator, should be excluded
* Patient has a least one measurable or assessable lesion according to RECIST 1.1 remaining after tumor resection for CC-38 manufacturing has been performed.
* Patient has ECOG performance status of 0 or 1.
* Patient has a minimum life expectancy of 6 months in the opinion of the investigator from the time of consent date.
* Patient has adequate bone marrow, hepatic and renal function in the opinion of the investigator:

  1. Hemoglobin ≥ 9.0 g/dL,
  2. Absolute neutrophil count (ANC) ≥ 1.0 x 109 /L,
  3. Platelets ≥ 80 x 109 /L,
  4. Calculated creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula),
  5. Serum bilirubin ≤ 1.5 x ULN (or ≤ 2.5 x ULN in the presence of documented Gilbert's Syndrome [unconjugated hyperbilirubinemia] or liver metastases),
  6. AST/ ALT and alkaline phosphatase ≤ 2.5 x ULN (or ≤5 times ULN in the presence of bone and/or liver metastases), ALP ≤ 2.5 x ULN,
  7. International normalized ration (INR) ≤ 1.5 or prothrombin time (PT) ≤ ULN + 4 seconds.
* Female patients must be post-menopausal or use contraceptive methods with a failure rate of < 1% 6 months after last administration of CC-38, whatever is later, to prevent pregnancy. Male patients with fertile female partners must be willing to use condoms with spermicide, and the fertile partner must use contraceptive methods with a failure rate of < 1% for the same time period. Male patients must also refrain from donating sperm for the same time period.
* Successful tumor tissue sampling by surgery, including presence of TILs in the tumor tissue in the pathological evaluation.
* Successful TIL expansion defined as obtaining the final CC-38 drug product

Exclusion Criteria:

* Patient as any of the following condition:

  1. Congestive heart failure NYHA class III or IV,
  2. myocardial infarction or coronary artery bypass graft within 6 months prior to enrollment,
  3. history of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration,
  4. history of severe non-ischemic cardiomyopathy,
  5. uncontrolled blood pressure as defined as systolic > 160 mmHg, diastolic > 100 mmHg within 3 months prior to enrollment,
  6. left ventricular ejection fraction (LVEF) < 45% as assessed by echocardiogram or multiple-gated acquisition (MUGA) scan,
  7. any other clinically significant cardiovascular events such as unstable angina, angioplasty, stroke, or transient ischemic attack (TIA) within less than 6 months before enrolment,
  8. other conditions that the treating physicians believe may endanger the health of the patients by their participation in this clinical trial.
* Patient has any of the following pulmonary conditions:

  1. Forced expiratory volume in 1 second (FEV1)<60%,
  2. Active obstructive chronic pulmonary disease,
  3. oxygen dependence as defined by a blood oxygen saturation that can only be maintained above 92% by oxygen inhalation (finger oxygen detection method),
  4. other pulmonary conditions that increase the anesthesiologic risk.
* Patient has a current or history of central nervous system (CNS) metastatic disease, leptomeningeal disease, or cord compression,
* Patient has ulcers in the upper GI tract, untreated or incompletely treated esophageal varices with high risk of bleeding in the investigator's discretion.
* Patient requiring therapeutic anticoagulant therapy or having other increased risk of bleeding events.
* Patient has any severe acute or chronic medical condition that places the patient at increased risk or interferes with the interpretation of trial results in the opinion of the investigator.
* Patient has any form of primary immunodeficiency (such as severe combined immunodeficiency disease [SCID] and acquired immune deficiency syndrome [AIDS]).
* Patient has active or history of autoimmune or inflammatory disorders. Note: Patients may be eligible if they have been assessed in discussion between Principal Investigator, Chief Medical Officer and Senior Medical Consultant as not posing an increased risk to the patient.
* Patient receiving immunosuppressive concomitant medications (≥ 10 mg prednisone daily or other equivalent). Steroid medications are allowed if they are used as substitution or are administrated topically or as inhalations.
* Patient has received an organ and/or allogenic stem cell transplant.
* Patient has known acute or chronic infection with hepatitis B or C virus.
* Patient has known HIV infection (seropositive for HIV antibody).
* Patient has known infection with syphilis.
* Patient has known bone-marrow aplasia.
* Patient has known (chronical) urinary tract infection and/ or acute urothelial toxicity from previous cytotoxic chemotherapy or radiation therapy or urinary flow obstructions.
* Female patient, who is pregnant or breast-feeding, or plan to become pregnant within 12 months after cyclophosphamide or 6 months after last dose of CC-38, whichever last. Women of childbearing potential must have a negative pregnancy test at screening and before every CC-38 application.
* Patient is unable to comply with trial procedures, restrictions, or requirements.
* Patient received last previous systemic cancer treatment (including anti-testosterone treatment) within less than 4 weeks prior enrollment.

Note: Bridging therapies (specified in trial design [section 2 - subsection: screening and TIL harvesting]) after TIL harvesting and before CC-38 administration are permitted after consultation between Principal Investigator, Chief Medical Officer and Senior Medical Consultant.

* Patient received last palliative radiotherapy within less than 4 weeks prior enrollment - where RECIST 1.1 evaluable metastases are within the radiation area.
* Patient received minor surgery (as judged by the investigator, i.e., port implantation) within less than 3 weeks prior enrollment.
* Patient with AEs from previous treatment that have not recovered to CTCAE v5.0 ≤ grade 1 Note: Clinically insignificant grade 2 AEs that may be allowable if discussed between and approved by Principal Investigator, Chief Medical Officer and Senior Medical Consultant.
* Patient participates in any other interventional clinical trial or has been treated with any investigational research products within 4 weeks prior to the initiation of screening.
* Patient has bone metastasis only.
* Patient has known hypersensitivity to any component of the trial regimen.
* For colorectal cancer: Patient has been diagnosed with histologically or cytologically proven BRAF-V600 positive CRC.
* Patient has any further contraindication to the IMP pembrolizumab or any of the auxiliary medicinal products (i.e., IL-2, cyclophosphamide, uromitexan) as per current EU SmPCs to the respective product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety, tolerability, and feasibility of repeated administrations of the novel ATIMP, CC-38. | 42 months
  Incidence of treatment-emerged adverse events (TEAE) and the occurrence of severity grade 3 or higher adverse events according to NCI CTCAE v. 5.0; proportion of patient receiving at least two CC-38 administrations without TEAEs preventing CC-38 administrations

SECONDARY OUTCOMES:
Evaluation of efficacy of repeated administrations of the novel ATIMP CC-38 in patients | 42 months
  Measurable objective response rate: Proportion of patients with complete [CR] or partial response [PR] as best response to treatment within the first 6 months after start of CC-38 administration (RECIST 1.1/iRECIST), or death from any cause, whichever comes first.
  Progression-free survival: time from start of treatment to time of disease progression (RECIST 1.1/ iRECIST), or death from any cause, whichever comes first.
  Time to tumor progression: time from start of treatment to disease progression (RECIST 1.1/iRECIST) Overall survival (OS): time from start of treatment to time of death from any cause.
  For prostate cancer cohort: Patient individual changes in prostate-specific antigen levels from baseline until 6 months after start of treatment.
  For colorectal cancer cohort: Patient individual changes in carcinoembryonic antigen and cancer antigen 19-9 levels from baseline until 6 months after start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Strom, Study Chair — Curacell Holding AB
Locations (1):
- Krankenhaus Nordwest, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No